CLINICAL TRIAL: NCT02152124
Title: Growth Hormone, IGF-1 and Medical Treatment in Acromegaly: Are There Effects on Gut Hormone Physiology and Postprandial Substrate Metabolism?
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: EC/2013/857; WI182140 (Other Grant/Funding Number: Pfizer)
Record Dates: First submitted 2014-05-21; First posted 2014-06-02 (Estimated); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Acromegaly
Keywords: Acromegaly; Acromegaly treatment; Long-acting somatostatin analogs; Pegvisomant; Insulin sensitivity; Gut hormones; Lipid metabolism; Adipokines
MeSH Terms: conditions — Acromegaly; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Controlled on LA-SMSA: Patients with controlled acromegaly on long-acting somatostatin analogs
- Controlled on LA-SMSA and pegvisomant: Patients with controlled acromegaly on long-acting somatostatin analogs and pegvisomant
- Controlled after surgery: Controlled acromegaly patients without need for medical therapy after surgery
- Healhy controls: Healthy volunteers
- Uncontrolled on LA-SMSA: Patients with uncontrolled acromegaly (i.e. with serum IGF-1 levels above age-specific thresholds and/or symptoms due to active acromegaly (e.g. excessive sweating, arthralgia)) on LA-SMSA monotherapy in maximal dosage

SUMMARY:
Acromegaly is a rare hormonal disorder leading to increased morbidity and mortality. In the vast majority of cases, a pituitary somatotroph cell adenoma causes excess growth hormone (GH) secretion, leading to hepatic insulin-like-growth factor 1 (IGF-1) hypersecretion. Both the disease as well as its treatment with long-acting somatostatin analogs (LA-SMSA) and/or pegvisomant affect glucose and lipid metabolism, possibly contributing to increased cardiovascular risk.

In this pilot study, the investigators want to explore insulin sensitivity, postprandial gut hormone response, lipid handling and adipocytokine profile in the following 4 groups:

* controlled acromegalic patients on LA-SMSA (group 1)
* controlled acromegalic patients on combination treatment of LA-SMSA and pegvisomant (group 2)
* acromegalic patients without need for medical therapy after surgery (group 3)
* healthy control subjects (group 4)

Furthermore, a longitudinal exploration will be performed in uncontrolled acromegalic patients (i.e. patients with serum IGF-1 levels above age-specific thresholds and/or symptoms due to active acromegaly (excessive sweating , arthralgia)) on LA-SMSA monotherapy (group 5). In this group, insulin sensitivity, postprandial gut hormone response, lipid handling and adipocytokine profile will be explored before introducing pegvisomant and three months after normalisation of IGF-1 levels.

The investigators hypothesize that lipid and glucose handling will be less efficient in the controlled acromegalic patients on LA-SMSA than in controlled patients on combination therapy or after surgery, and that there will be no difference in substrate metabolism between healthy controls and controlled acromegalic patients on combination treatment or after surgery. Further, they hypothesize that introducing pegvisomant in uncontrolled acromegalic patients will improve their postprandial lipid and glucose handling.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acromegaly over 1 year ago, no changes in treatment schedule since at least 6 months (groups 1-3 and 5) OR healthy volunteer without diagnosis of acromegaly (group 4)
* Patient is willing to participate and has signed the informed consent
* Age > 18 years and < 80 years
* Body Mass Index 18-40 kg/m²

Exclusion Criteria:

* Biochemistry: liver function tests > 3x ULN; HbA1C > 58 mmol/mol
* All untreated endocrine disorders including uncontrolled diabetes mellitus type 2 (i.e. HbA1C > 58 mmol/mol)
* Bariatric surgery; malabsorptive syndromes; hepatic or renal failure
* Current medication use: insulin, metformin, sulfonylurea, fibrates, incretin mimetics, dopamine agonists (for all but insulin, participation is allowed after a 2- week wash-out period)
* Abuse of alcohol or drugs
* Weight changes > 10% of body weight during preceding 12 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Groups 1-3 and 5: outpatient clinic attendants Group 4: recruted from community (by placard)
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
change in insulin sensitivity | before start of pegvisomant and 3 months after normalisation of IGF-1 after start of pegvisomant in group 5
  Glucose disposal rate during last half hour of hyperinsulinemic-euglycemic clamp procedure, corrected for lean body mass (in µmol/min/kgLBM)
insulin sensitivity | At enrollment in groups 1-4
  Glucose disposal rate during last half hour of hyperinsulinemic-euglycemic clamp procedure, corrected for lean body mass (in µmol/min/kgLBM)

SECONDARY OUTCOMES:
fasting and postprandial glucose | At enrollment in groups 1-4
  Serum glucose levels during mixed-meal test (before and 10, 30, 60, 120, 180, 240, 300 minutes after ingestion of standard mixed-meal (bread, margarine, cheese and milk) providing a caloric content of 1000 kCal whereby 45% of the energy comes from fat, 36% from carbohydrates and 19% from proteins)
fasting and postprandial insulin | At enrollment in groups 1-4
  Insulin levels during standard mixed-meal test (cfr.supra)
fasting and postprandial gut hormone levels | At enrollment in groups 1-4
  Serum levels of gastric inhibitory polypeptide (GIP), ghrelin, peptide YY, pancreatic polypeptide, glucagon-like peptide 1 (GLP-1), oxyntomodulin and cholecystokinin before start during standard mixed-meal test (cfr.supra)
fasting adipokine levels | At enrollment in group 1-4
  Fasting serum levels of leptin, adiponectin and interleukin 6 (IL-6)
fasting lipid levels | At enrollment in groups 1-4
  Fasting serum levels of triglycerides, total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol
change in fasting and postprandial glucose | before start of pegvisomant and 3 months after normalisation of IGF-1 levels after start of pegvisomant in group 5
  Serum glucose levels during mixed-meal test (before and 10, 30, 60, 120, 180, 240, 300 minutes after ingestion of standard mixed-meal (bread, margarine, cheese and milk) providing a caloric content of 1000 kCal whereby 45% of the energy comes from fat, 36% from carbohydrates and 19% from proteins)
change in fasting and postprandial insulin levels | before start of pegvisomant and 3 months after normalisation of IGF-1 levels after start of pegvisomant in group 5
  Insulin levels during standard mixed-meal test (cfr.supra)
change in fasting and postprandial gut hormone levels | before start of pegvisomant and 3 months after normalisation of IGF-1 levels after start of pegvisomant in group 5
  Serum levels of gastric inhibitory polypeptide (GIP), ghrelin, peptide YY, pancreatic polypeptide, glucagon-like peptide 1 (GLP-1), oxyntomodulin and cholecystokinin before start during standard mixed-meal test (cfr.supra)
change in fasting adipokine levels | before start of pegvisomant and 3 months after normalisation of IGF-1 levels after start of pegvisomant in group 5
  Fasting serum levels of leptin, adiponectin and interleukin 6 (IL-6)
change in fasting lipid levels | before start of pegvisomant and 3 months after normalisation of IGF-1 levels after start of pegvisomant in group 5
  Fasting serum levels of triglycerides, total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol

OTHER OUTCOMES:
Resting energy expenditure | At enrollment in group 1-4
  Resting energy expenditure determined using indirect calorimetry
Weight | At enrollment in group 1-4
Standing height | At enrollment in group 1-4
Waist and hip circumference | At enrollment in group 1-4
Change in resting energy expenditure | before start of pegvisomant and 3 months after normalisation of IGF-1 levels after start of pegvisomant in group 5
  Resting energy expenditure determined using indirect calorimetry
Weight change | before start of pegvisomant and 3 months after normalisation of IGF-1 levels after start of pegvisomant in group 5
Change in standing height | before start of pegvisomant and 3 months after normalisation of IGF-1 levels after start of pegvisomant in group 5
Change in waist and hip circumference | before start of pegvisomant and 3 months after normalisation of IGF-1 levels after start of pegvisomant in group 5

CONTACTS AND LOCATIONS:
Overall Officials: Guy T'Sjoen, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Department of Endocrinology, 9K12IE, Ghent, Belgium

REFERENCES:
- [Background] Baldelli R, Battista C, Leonetti F, Ghiggi MR, Ribaudo MC, Paoloni A, D'Amico E, Ferretti E, Baratta R, Liuzzi A, Trischitta V, Tamburrano G. Glucose homeostasis in acromegaly: effects of long-acting somatostatin analogues treatment. Clin Endocrinol (Oxf). 2003 Oct;59(4):492-9. doi: 10.1046/j.1365-2265.2003.01876.x. PMID 14510913
- [Background] Barkan AL, Burman P, Clemmons DR, Drake WM, Gagel RF, Harris PE, Trainer PJ, van der Lely AJ, Vance ML. Glucose homeostasis and safety in patients with acromegaly converted from long-acting octreotide to pegvisomant. J Clin Endocrinol Metab. 2005 Oct;90(10):5684-91. doi: 10.1210/jc.2005-0331. Epub 2005 Aug 2. PMID 16076947
- [Background] Berg C, Petersenn S, Lahner H, Herrmann BL, Buchfelder M, Droste M, Stalla GK, Strasburger CJ, Roggenbuck U, Lehmann N, Moebus S, Jockel KH, Mohlenkamp S, Erbel R, Saller B, Mann K; Investigative Group of the Heinz Nixdorf Recall Study and the German Pegvisomant Observational Study Board and Investigators. Cardiovascular risk factors in patients with uncontrolled and long-term acromegaly: comparison with matched data from the general population and the effect of disease control. J Clin Endocrinol Metab. 2010 Aug;95(8):3648-56. doi: 10.1210/jc.2009-2570. Epub 2010 May 12. PMID 20463098
- [Background] Colao A, Pivonello R, Auriemma RS, De Martino MC, Bidlingmaier M, Briganti F, Tortora F, Burman P, Kourides IA, Strasburger CJ, Lombardi G. Efficacy of 12-month treatment with the GH receptor antagonist pegvisomant in patients with acromegaly resistant to long-term, high-dose somatostatin analog treatment: effect on IGF-I levels, tumor mass, hypertension and glucose tolerance. Eur J Endocrinol. 2006 Mar;154(3):467-77. doi: 10.1530/eje.1.02112. PMID 16498061
- [Background] De Marinis L, Bianchi A, Fusco A, Cimino V, Mormando M, Tilaro L, Mazziotti G, Pontecorvi A, Giustina A. Long-term effects of the combination of pegvisomant with somatostatin analogs (SSA) on glucose homeostasis in non-diabetic patients with active acromegaly partially resistant to SSA. Pituitary. 2007;10(3):227-32. doi: 10.1007/s11102-007-0037-7. PMID 17484056
- [Background] Freda PU, Reyes CM, Conwell IM, Sundeen RE, Wardlaw SL. Serum ghrelin levels in acromegaly: effects of surgical and long-acting octreotide therapy. J Clin Endocrinol Metab. 2003 May;88(5):2037-44. doi: 10.1210/jc.2002-021683. PMID 12727951
- [Background] Kim SK, Suh S, Lee JI, Hur KY, Chung JH, Lee MK, Min YK, Kim JH, Kim JH, Kim KW. The ability of beta-cells to compensate for insulin resistance is restored with a reduction in excess growth hormone in Korean acromegalic patients. J Korean Med Sci. 2012 Feb;27(2):177-83. doi: 10.3346/jkms.2012.27.2.177. Epub 2012 Jan 27. PMID 22323865
- [Background] Kozakowski J, Rabijewski M, Zgliczynski W. [Lowered ghrelin levels in acromegaly-normalization after treatment]. Endokrynol Pol. 2005 Nov-Dec;56(6):862-70. Polish. PMID 16821203
- [Background] Mazziotti G, Floriani I, Bonadonna S, Torri V, Chanson P, Giustina A. Effects of somatostatin analogs on glucose homeostasis: a metaanalysis of acromegaly studies. J Clin Endocrinol Metab. 2009 May;94(5):1500-8. doi: 10.1210/jc.2008-2332. Epub 2009 Feb 10. PMID 19208728
- [Background] Moller N, Jorgensen JO. Effects of growth hormone on glucose, lipid, and protein metabolism in human subjects. Endocr Rev. 2009 Apr;30(2):152-77. doi: 10.1210/er.2008-0027. Epub 2009 Feb 24. PMID 19240267
- [Background] Moller L, Norrelund H, Jessen N, Flyvbjerg A, Pedersen SB, Gaylinn BD, Liu J, Thorner MO, Moller N, Lunde Jorgensen JO. Impact of growth hormone receptor blockade on substrate metabolism during fasting in healthy subjects. J Clin Endocrinol Metab. 2009 Nov;94(11):4524-32. doi: 10.1210/jc.2009-0381. Epub 2009 Oct 9. PMID 19820031
- [Background] Neggers SJ, Kopchick JJ, Jorgensen JO, van der Lely AJ. Hypothesis: Extra-hepatic acromegaly: a new paradigm? Eur J Endocrinol. 2011 Jan;164(1):11-6. doi: 10.1530/EJE-10-0969. Epub 2010 Nov 2. PMID 21045065
- [Background] Peracchi M, Porretti S, Gebbia C, Pagliari C, Bucciarelli P, Epaminonda P, Manenti S, Arosio M. Increased glucose-dependent insulinotropic polypeptide (GIP) secretion in acromegaly. Eur J Endocrinol. 2001 Jul;145(1):R1-4. doi: 10.1530/eje.0.145r001. PMID 11415859
- [Background] Pierluissi J, de Pierluissi RM. Effect of glucose-dependent insulinotropic polypeptide (GIP) on insulin response to glucose in acromegalics. Acta Cient Venez. 1995;46(2):89-96. PMID 9279024
- [Background] Plockinger U, Holst JJ, Messerschmidt D, Hopfenmuller W, Quabbe HJ. Octreotide suppresses the incretin glucagon-like peptide (7-36) amide in patients with acromegaly or clinically nonfunctioning pituitary tumors and in healthy subjects. Eur J Endocrinol. 1999 Jun;140(6):538-44. doi: 10.1530/eje.0.1400538. PMID 10377503
- [Background] Velasquez-Mieyer PA, Umpierrez GE, Lustig RH, Cashion AK, Cowan PA, Christensen M, Spencer KA, Burghen GA. Race affects insulin and GLP-1 secretion and response to a long-acting somatostatin analogue in obese adults. Int J Obes Relat Metab Disord. 2004 Feb;28(2):330-3. doi: 10.1038/sj.ijo.0802561. PMID 14708034